CLINICAL TRIAL: NCT07035756
Title: Development of an Arterial Pressure Monitoring Set Fixation Apparatus and Evaluation of Its Effectiveness
Brief Title: Development of an Arterial Pressure Monitoring Set Fixation Apparatus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Zeynep Gürkan, Research Assistant and PhD Candidate, Yuzuncu Yil University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2024/08-09; TDK-2024-14774 (Other Grant/Funding Number: Atatürk Univ. Sci. Res. Projects Coord. Unit)
Record Dates: First submitted 2025-06-12; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: Arterial Pressure Monitoring; Fixation Device; Coronary Artery Bypass Graft (CABG); Hemodynamic Monitoring; Postoperative Care

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled sequentially and receive the new arterial pressure monitoring set fixation device. Data on fixation stability, patient comfort, and hemodynamic parameters will be collected over 48 hours postoperatively to assess the device's performance.
Masking Description: The study is not blinded; participants and investigators know which intervention is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arterial Pressure Monitoring Set Fixation Device Group (Experimental): This group includes patients who will receive the new arterial pressure monitoring set fixation device. The device is applied postoperatively to secure arterial pressure monitoring and improve fixation stability and patient comfort over a 48-hour period.
  Interventions: Device: Arterial Pressure Monitoring Set Fixation Device

INTERVENTIONS:
Device: Arterial Pressure Monitoring Set Fixation Device — A newly developed fixation device designed to securely stabilize the arterial pressure monitoring set, improving patient comfort and reducing device displacement during the postoperative period in patients undergoing coronary artery bypass graft surgery.

SUMMARY:
This study aims to develop an arterial pressure monitoring set fixation device and evaluate its effectiveness in clinical settings. The device is designed to increase the stability and comfort of arterial pressure monitoring during patient care. An experimental study will be conducted with patients requiring arterial pressure monitoring. The device's effectiveness will be evaluated by measuring fixation stability and postoperative arterial blood pressure-CVP parameters over 48 hours. The study aims to demonstrate that the new fixation device can improve patient safety and monitoring accuracy compared to the standard method using adhesive tape, thereby contributing to better clinical outcomes.

DETAILED DESCRIPTION:
This study focuses on the development of a novel arterial pressure monitoring set fixation device designed to enhance stability and comfort during invasive arterial pressure measurement. The device securely fixes the monitoring set in place, reducing movement and potential complications caused by displacement or discomfort associated with the adhesive tapes currently in use.

An experimental study design will be employed. Sixty patients requiring postoperative invasive arterial pressure monitoring will be included based on predefined inclusion and exclusion criteria. The fixation device will be applied to these patients.

Fixation stability, patient comfort, and hemodynamic parameters, including arterial blood pressure and central venous pressure (CVP), will be measured over a 48-hour postoperative period. The data will be analyzed to evaluate the device's effectiveness in improving monitoring accuracy and patient safety.

Ethical approval has been obtained from the relevant institutional review board, and compliance with human subject protection standards will be maintained throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-80 years
* Patients undergoing arterial catheterization for invasive blood pressure and CVP monitoring
* Patients able to provide informed consent
* Hemodynamically stable patients undergoing Coronary Artery Bypass Grafting (CABG)

Exclusion Criteria:

* Patients younger than 18 or older than 80 years
* Patients with coagulopathy or bleeding disorders
* Patients with local infection or skin lesions at the catheter insertion site
* Patients unable to provide informed consent
* Hemodynamically unstable patients
* Patients with known allergy to device materials or adhesive tapes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Invasive Blood Pressure and Central Venous Pressure Measurements | Within the first 48 hours of monitoring
  The accuracy of arterial and central venous pressure measurements obtained using the developed fixation device will be compared to those obtained using standard adhesive tape fixation. Accuracy will be determined by evaluating waveform stability and consistency of numeric readings during patient movement and routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Gürkan, Res. Asst., Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van Training and Research Hospital, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Result] Nguyen Y, Bora V. Arterial Pressure Monitoring. 2023 Mar 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK556127/ PMID 32310587